CLINICAL TRIAL: NCT05957926
Title: Evaluation the Effect of Hyaluronic Acid With Hydroxyapatite Versus Hydroxyapatite Alone on Bone Regeneration Following Enucleation of Mandibular Odontogenic Cyst (Randomized Clinical Trial)
Brief Title: Hyaluronic Acid +Hydroxyapatite Vs Hydroxyapatite in Bone Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas Fadel Said Aldaour, Bachelor of Dental Surgery ( BDS ), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2991
Record Dates: First submitted 2023-07-08; First posted 2023-07-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-07

CONDITIONS: Bone Loss; Bone Lesion
Keywords: bone regenerarion; bone graft; hydroxyapatite
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Durapatite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid + Hydroxyapatite (Experimental): hyaluronic acid is used for bone regeneration and it has a good potential for osteogenesis and mineralization so it can have synergistic effect when used with hydroxyapatite for bone regeneration after cyst enucleation
  Interventions: Procedure: hyaluronic acid added to hydroxyapetite
- Hydroxyapatite alone (Active Comparator): Hydroxyapatite is inorganic component of bone tissue used as bone graft, scaffolds, filler and cement for repair and regeneration of bone defect , and it stimulates bone remodeling by generating surface active moieties or cell signaling process
  Interventions: Procedure: Hydroxyapatite alone

INTERVENTIONS:
Procedure: hyaluronic acid added to hydroxyapetite — 1. The procedure will be performed under complete aseptic condition, and the surgical field will be swabbed with povidone iodine solution before the operation .
  2. Surgical procedure will be performed under local anesthesia (Articaine 4% with 1:100,000 adrenaline ) .
  3. A full thickness mucoperiosteal flap will be reflected exposing the area of interest containing the lesion .
  4. The pathological lesion will be exposed using rose head bur on low-speed handpiece under copious irrigation by normal saline .
  5. The whole pathological tissues will be enucleated and sent for histopathological examination.
  6. The cavity will be curetted again to remove any remaining tissues and irrigated with 0.9% normal saline .
  7. hydroxyapetite with hyaluronic acid will be inserted in the bony cavity to initiate healing .
  8. The flap will be repositioned and sutured with interrupted 3-0 Vicryl suture .
  Arms: Hyaluronic acid + Hydroxyapatite
Procedure: Hydroxyapatite alone — 1. The procedure will be performed under complete aseptic condition, and the surgical field will be swabbed with povidone iodine solution before the operation .
  2. Surgical procedure will be performed under local anesthesia (Articaine 4% with 1:100,000 adrenaline ) .
  3. A full thickness mucoperiosteal flap will be reflected exposing the area of interest containing the lesion .
  4. The pathological lesion will be exposed using rose head bur on low-speed handpiece under copious irrigation by normal saline .
  5. The whole pathological tissues will be enucleated and sent for histopathological examination.
  6. The cavity will be curetted again to remove any remaining tissues and irrigated with 0.9% normal saline .
  7. hydroxyapetite will be inserted in the bony cavity to initiate healing .
  8. The flap will be repositioned and sutured with interrupted 3-0 Vicryl suture .
  Arms: Hydroxyapatite alone

SUMMARY:
Evaluation of the effect of hyaluronic acid with hydroxyapatite versus hydroxyapatite alone on bone regeneration following enucleation of mandibular odontogenic cyst.

DETAILED DESCRIPTION:
During cyst enucleation , There's resultant decrease in bone density especially in large defects .Therefore, it may be needed for a bone grafts and bone regenerative materials to improve quality of bone .The rationale is to evaluate hyaluronic acid with hydroxyapatite as a bone quality improvement material following cyst enucleation, which would provide significant bone regeneration. Hydroxyapatite is inorganic component of bone tissue used as bone graft, scaffolds, filler and cement for repair and regeneration of bone defect , and it is stimulate bone remodeling by generating surface active moieties or cell signaling process while Hyaluronic acid and it's derivatives has been widely used for bone regeneration and it has a good potential for osteogenesis and mineralization

ELIGIBILITY:
Inclusion Criteria:

* Patient in need of cyst removal .
* Both genders aged between 18-50 years .
* Size of lesion is ≤ 4 cm .
* Patients free from any systemic disease that may affect bone healing .

Exclusion criteria :

* Heavy smokers , alcohol intake .
* Poor oral hygiene .
* Patient with systemic disease that may affect bone healing .
* Pregnant women.
* Patient who are currently or have been under treatment using chemotherapy or radiotherapy
* Uncooperative patient .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Bone density | 6 months
  It is assessed using CBCT to determine the density of bone after intervention

SECONDARY OUTCOMES:
postoperative pain | 2 weeks
  It is assessed by using visual analogue scale from 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao N, Wang X, Qin L, Zhai M, Yuan J, Chen J, Li D. Effect of hyaluronic acid in bone formation and its applications in dentistry. J Biomed Mater Res A. 2016 Jun;104(6):1560-9. doi: 10.1002/jbm.a.35681. Epub 2016 Apr 9. PMID 27007721
- [Background] Scariot R, da Costa DJ, Rebellato NL, Muller PR, Gugisch RC. Treatment of a large dentigerous cyst in a child. J Dent Child (Chic). 2011 Jul;78(2):111-4. PMID 22041117
- [Background] AboulHosn M, Noujeim Z, Nader N, Berberi A. Decompression and Enucleation of a Mandibular Radicular Cyst, Followed by Bone Regeneration and Implant-Supported Dental Restoration. Case Rep Dent. 2019 Jan 9;2019:9584235. doi: 10.1155/2019/9584235. eCollection 2019. PMID 30729045